CLINICAL TRIAL: NCT00984516
Title: A Single-site, Placebo-controlled, Double-blind Trial to Investigate the Safety, Tolerability, Systemic Exposure and the Scar-improvement Efficacy of Intradermal Applications of Three Doses of Juvidex (5.64mg/100μl, 2.82mg/100μl and 11.28mg/100μl) Given Once Only or Three Times Within and Between Male and Female Subjects Aged 18-45.
Brief Title: Investigation Into the Safety and Scar-improvement Efficacy of Intradermal Juvidex Dosed Once or Three Times
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Medical Director, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1004-319-1002
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound-healing
Keywords: Cicatrix; Scar; Wound-healing; Juvidex; Mannose-6-phosphate; M6P; RN1004
MeSH Terms: conditions — Cicatrix | interventions — mannose-6-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal Juvidex (Experimental)
  Interventions: Drug: Juvidex
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Juvidex — Intradermal Juvidex, 100μl of 100mM (2.82mg/100μl) administered once prior to wounding
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 100mM (2.82mg/100μl) administered once prior to wounding, once 3 hours later at 100μl/wound margin (200μl total) and again on Day 5 (200μl)
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 200mM (5.64mg/100μl) administered once prior to wounding
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 200mM (5.64mg/100μl) administered once prior to wounding, once 3 hours later at 100μl/wound margin (200μl total) and again on Day 5 (200μl)
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 400mM (11.28mg/100μl) administered once prior to wounding
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 400mM (11.28mg/100μl) administered once prior to wounding, once 3 hours later at 100μl/wound margin (200μl total) and again on Day 5 (200μl)
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Placebo — Intradermal Placebo, 100μl administered once prior to wounding
  Arms: Placebo (vehicle)
Drug: Placebo — Intradermal Placebo, 100μl administered once prior to wounding, once 3 hours later at 100μl/wound margin (200μl total) and again on Day 5 (200μl)
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study was to investigate the scar-improvement efficacy of three doses of intradermal Juvidex given once only or three times in male and female subjects and to collect further safety and tolerability data for intradermal Juvidex in male and female subjects.

DETAILED DESCRIPTION:
Subjects were randomised into three dose groups of equal size. The three dose groups were 100mM (2.82mg/100μl), 200mM (5.64mg/100μl) and 400mM (11.28mg/100μl). Before wounding, three prospective wound sites 1cm long were marked on the upper, inner aspect of each arm (anterior, posterior and distal) to give three pairs of wounds. Wounds were assigned as Pair 1 (left distal and right distal), Pair 2 (left anterior and left posterior) and Pair 3 (right anterior and right posterior).

Sites were anaesthetised using 1% plain lignocaine, then prior to wounding one site from each pair, randomly assigned, received an intradermal injection of Juvidex (100μl) and the opposite site from each pair received an intradermal injection of Placebo (100μl).

Within dose groups, subjects were randomised into two subgroups of similar size. Subgroup A received one dose in wound pairs 1 and 2; and three doses in wound pair 3. Subgroup B received three doses in wound pairs 1 and 2; and one dose in wound pair 3. Incision sites randomised to receive three injections of study medication were re-dosed with 100μl per wound margin (200μl per site) 3 hours after receiving the first dose and dosed again in the same way on Day 5.

Subjects attended a follow-up visit on Day 14. Scars were assessed monthly from Month 1 to Month 12. At Month 12, the Investigator excised the distal scars from each subject for histological examination. Posttrial follow-up visits are scheduled for Months 18 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-45 years who gave written informed consent
* Weight between 50-150kg with a BMI within the permitted range for their height using Quetelet's index: weight (kg)/height (m)2. The permitted range was 15-55kg/m2
* Female subjects of childbearing potential who were deemed by the Investigator to be using adequate contraception at the time of screening and who agreed to continue using this form of contraception for the duration of the trial
* In the opinion of the Investigator, and on the basis of the investigations carried out within 12 weeks prior to the first study drug dose (determined by results of electrocardiogram [ECG], physical examination, medical history, haematology and biochemistry blood results) the subject was in adequate health to undertake the trial

Exclusion Criteria:

* Subjects who on direct questioning and physical examination had a history or evidence of hypertrophic or keloid scarring or had tattoos in the area to be incised
* Afro-Caribbean subjects because of their increased susceptibility to hypertrophic and keloid scarring
* Subjects who had surgery in the area to be incised within one year of the first dosing day
* Subjects with a history of a bleeding disorder
* Subjects who, on direct questioning and physical examination, had evidence of any past or present clinically significant disease, particularly coagulation disorders, diabetes, immuno-mediated conditions and skin diseases and allergies, such as clinically significant eczema
* Subjects with a skin disorder that was chronic or currently active and which the Investigator considered would adversely affect the healing of the acute wounds or would involve the areas to be examined in this trial
* Subjects with any clinically significant medical condition that would impair wound healing including; significant rheumatoid arthritis, chronic renal impairment significant for their age, significant hepatic impairment (LFTs >3 times upper limit of normal), congestive heart failure, current active malignancy or history of malignancy in the last 5 years, immunosuppression or chemotherapy within the last 12 months, a history of radiotherapy and diabetes mellitus
* Subjects with a history of clinically significant drug hypersensitivity to lignocaine or an allergy to surgical dressings to be used in this trial
* Subjects who were taking or had taken any investigational product or participated in a clinical trial within the three months prior to first study drug dose for this trial
* Subjects who were taking regular, continuous, oral corticosteroid therapy
* Subjects who, in the opinion of the Investigator, were not likely to complete the trial for whatever reason
* Subjects who were, or who became, pregnant or were lactating, up to and including the time of the first dose of study drug
* Subjects undergoing/awaiting investigations or change in management for an existing medical disorder
* Subjects who had evidence of drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To investigate the scar-improvement efficacy of three doses of intradermal Juvidex given once only and three times in male and female subjects. | 12 months

SECONDARY OUTCOMES:
To collect further safety and tolerability data for various doses and dosing frequencies of intradermal Juvidex in male and female subjects. | 1 hour to 24 months
To assess systemic exposure to Juvidex, following various doses and dosing frequencies of intradermal Juvidex, before and after making minor skin incisions in male and female subjects. | 1 hour to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Bush, Principal Investigator — Renovo
Locations (1):
- Renovo, Manchester, United Kingdom